CLINICAL TRIAL: NCT02082899
Title: A Single Center, Randomized, Double-Masked, Vehicle-Controlled, Parallel, Group Study to Assess the Efficacy of EBI-005 Topical Ophthalmic Solution for the Treatment of Moderate to Severe Allergic Conjunctivitis Using an Environmental Exposure Chamber (EEC) Model and Conjunctival Allergen Provocation Test (CAPT) Model
Brief Title: A Single Center Study for the Treatment of Moderate to Severe Allergic Conjunctivitis (EBI-005-AC-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBI-005-AC-1
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic Conjunctivitis; Interleukin 1 Receptor Inhibitor; Environmental Exposure Chamber; Conjunctival Allergen Provocation Test
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator EBI-005 5 mg/mL (Active Comparator): Administered 3 times per day
  Interventions: Drug: Active Comparator EBI-005 5 mg/mL
- Placebo Comparator (Placebo Comparator): Administered 3 times per day
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Active Comparator EBI-005 5 mg/mL
  Arms: Active Comparator EBI-005 5 mg/mL
Drug: Placebo Comparator
  Arms: Placebo Comparator

SUMMARY:
This is a Phase II Single Center, Randomized, Double-Masked, Vehicle-Controlled, Parallel, Group Study to Assess the Efficacy of EBI-005 Topical Ophthalmic Solution for the Treatment of Moderate to Severe Allergic Conjunctivitis Using an Environmental Exposure Chamber (EEC) Model and Conjunctival Allergen Provocation Test (CAPT) Model. Approximately 150 subjects will be enrolled and randomized in one study center in Canada for a duration of 0.33 years.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to any study-related procedures.
* Be 18 years of age or older.
* Have at least a 2 year history of moderate to severe allergic conjunctivitis.
* Have a positive skin prick test to ragweed within the past 12 months of Screening (Visit 1A).
* Have a score of ≥ 2 for staff-assessed ocular redness in at least one region (nasal or temporal) in each eye and ≥ 2 for subject-assessed ocular itching within the 3.5-hour period of allergen exposure in the EEC at Visit 1B.
* Have required more than one anti-allergy pharmaceutical treatments in the past 2 years to treat ocular symptoms (including oral, topical, nasal treatments).
* Be able to self-administer topical ophthalmic drops.
* Avoid any topical or systemic ocular medications during the entire study period.
* Are willing and able to follow instructions and can be present for the required study visits for the duration of the study.

Exclusion Criteria:

* Are female and of childbearing potential and unwilling to remain abstinent through 30 days following the last dose of study drug or not willing to use acceptable birth control methods.
* Have previously used an IL-1 blocker (e.g., Anakinra, Rilonacept, or Ilaris).
* Have a known contraindication or hypersensitivities to Anakinra (Kineret®) or any therapeutic agent targeted to IL-1 or any component of study drug formulation.
* Current participation in another clinical study involving an experimental treatment or participation in such a study within 30 days prior to study entry.
* Require concomitant use of TNF-blocking agents (e.g., Etanercept, Adalimumab, Infliximab).
* Have a history of glaucoma or intraocular pressure (IOP) > 25 mmHg at the Visit 1A (Medical Screening) or a history of elevated IOP within the past year.
* Have had ocular surgery including laser procedures within the past 12 months of Visit 1A (Medical Screening).
* Have had contact lens wear within 4 weeks prior to Visit 1A (Medical Screening) or unwilling to discontinue wear during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Ocular itching in EEC arm at a specific visit comparing EBI-005 vs vehicle | 17 days

SECONDARY OUTCOMES:
Evaluation of Adverse Events. | up to 45 days
  Frequency, severity and relationship to study medication of all Adverse Events occurring during the study.
Evaluation of antibodies to EBI-005. | up to 45 days
  Number and percent of subjects who develop drug antibodies over time
Evaluation of ocular changes | up to 45 days
  Changes in ophthalmic examinations over time.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, MD, Study Director — Eleven Biotherapeutics
Locations (1):
- Investigation Site, Mississauga, Ontario, Canada